CLINICAL TRIAL: NCT04942405
Title: Efficacy, Immunogenicity, and Safety of the Two-Dose Inactivated COVID-19 Vaccine (TURKOVAC) Versus the Two-Dose CoronaVac (Sinovac) Vaccine in Healthy Subjects: A Randomized, Observer-Blinded, Phase III Clinical Trial
Brief Title: Efficacy, Immunogenicity, and Safety of the Inactivated COVID-19 Vaccine (TURKOVAC) Versus the CoronaVac Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TSB-VAC-COV-TUR-F3.01
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Covid19
Keywords: COVID-19, SARS-CoV-2 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TURKOVAC SARS-COV-2 Vaccine (Experimental): 600 Subunit of SARS-CoV-2 virus antigen, intramuscular injection, two doses given 28 days apart.
  Interventions: Biological: TURCOVAC
- CoronaVac (Active Comparator): 600 Subunit of SARS-CoV-2 virus antigen, intramuscular injection, two doses given 28 days apart.
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: TURCOVAC — Two doses at 28-day interval, each inoculation dose is 0.5 mL. Two doses of dosage (vaccine contains 600 subunit of SARS-CoV-2 virus antigen) experimental vaccine at the schedule of day 0,28
  Arms: TURKOVAC SARS-COV-2 Vaccine
Biological: CoronaVac — Two doses at 28-day interval, each inoculation dose is 0.5 mL. Two doses of dosage (vaccine contains 600 subunit of SARS-CoV-2 virus antigen) vaccine at the schedule of day 0, 28
  Arms: CoronaVac

SUMMARY:
This study is a randomized, double-blinded, and active-controlled phase III clinical trial of the SARS-CoV-2 inactivated vaccine. The purpose of this study is to evaluate the efficacy, safety, and immunogenicity of the experimental vaccine in healthy adults aged 18~55 years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, multi-center, active-controlled phase III clinical trial in adults aged 18~55 years. The purpose of this study is to evaluate the efficacy, safety, and immunogenicity of the experimental SARS-CoV-2 inactivated vaccine. A total of 40.800 subjects will be enrolled. The participant will be assigned to receive two doses of experimental vaccine or CoronaVac on the schedule of days 0, 28.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the following criteria to be enrolled in this study:

1. Subjects consented voluntarily to participate the study,
2. Subjects agreed to comply with all study visits and procedures (consented to give blood sample and nasopharyngeal swab, and receiving automated telephone calls from the study site),
3. Subjects agreed to adhere to the prohibitions and restrictions specified in this protocol,
4. Subjects, who are sexually active and have childbearing potential, agreed to comply with the contraceptive requirements to be applied in the study,
5. Adult males or females of at least 18 years of age and not older than 55 years of age on the date of the informed consent signature,
6. Subjects who are medically stable (those without severe pain, severe swelling, severe movement limitation, persistent high fever, severe headache or other systemic or local reactions) such that who are not anticipated to hospitalize within the study period, according to the judgment of the Investigator, and the subjects appears likely to be able to continue the study until the follow-up period specified in the protocol,
7. Subjects who are excluded from the criteria to receive the COVID-19 vaccine approved in the scope of Emergency Use Approval in Turkey or subjects who meet the vaccination criteria, but voluntarily chose not to be vaccinated and agreed to receive one of the vaccines to be used in this study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Is acutely ill or febrile within 48 hours before or use of antipyretic or analgesic medication within 24 hours before planned administration of study vaccine. (Fever is defined as a body temperature is 38.0 °C. Subjects with mild illness and fever may be enrolled in the study at the discretion of the investigator).
2. Subjects who are pregnant or breastfeeding.
3. Known history of SARS-CoV-2 infection.
4. Individuals with a current positive (PCR-based viral RNA detection) or past positive (serological testing or PCR-based viral RNA detection) diagnostic test result for SARS-CoV-2 infection.
5. Prior administration of an investigational or approved coronavirus (SARS-CoV, SARS-CoV-2, MERS-CoV) vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19.
6. Subjects determined as ineligible to the study protocol.
7. Subjects with a history of cardiac diseases (cardiovascular disease, serious arrythmia, coronary artery disease, heart failure, cardiomyopathies, pulmonary hypertension etc).
8. Subjects with uncontrolled hypertension.
9. Subjects with a family history of coronary artery disease at early ages (presence of before age 55 in men and before age 65 in women).
10. Subjects with morbid obesity (Body mass index (BMI) ≥ 40).
11. Subjects who have a travel plan to out of the city up to 28 days after the second vaccine dose.
12. Subjects with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and autoimmune bullous diseases.
13. Subjects with history of severe allergic reaction (i.e., anaphylaxis, generalized urticaria, angioedema, or other significant reaction) to any licensed or investigational vaccine or to any of the constituents of CoronaVac or TURKOVAC.
14. Subjects who has bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
15. Immunosuppressive or immunodeficient state (including HIV), asplenia, recurrent severe infections.
16. Subjects who have medical conditions that prioritize them for receipt of approved COVID-19 vaccine in Turkey and has a valid vaccination right within the Ministry of Health vaccination programme.
17. Subjects who received or planned to receive a licensed, live replicating vaccine (any vaccine other than the COVID-19 vaccine) within 28 days before or after first study vaccination or a licensed inactivated or non-replicating vaccine (any vaccine other than the COVID-19 vaccine) within 14 days before or after first study vaccination.
18. Subjects who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, e.g., for cancer or an autoimmune disease, within 6 months prior to screening, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study vaccine administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
19. Subjects who received systemic immunoglobulins or blood products within 3 months prior to the Day 0 or plans to receive such products during the study.
20. Investigator site staff members, employees of TUSEB or the Clinical Research Organization (CRO) directly involved in the conduct of the study, or site staff members otherwise supervised by the Investigator or immediate family members of any of the previously mentioned individuals.

Exclusion criteria for the second dose of vaccine:

1. Laboratory-confirmed SARS-CoV-2 infection after the first vaccination.
2. In case of an acute disease that has not recovered before the second vaccination or at acute phase of a chronic disease, the investigator should exclude COVID-19, and assess if the acute disease can recover in a short term.
3. New or newly occurred non-compliance with the inclusion/exclusion criteria after the first dose, which will be assessed by the investigator whether the study participation can continue or not.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1290 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Protection Indexes of Two Vaccine Doses For Symptomatic COVID-19. | 2 weeks after the second dose of vaccination
  To evaluate the efficacy of two-dose regimen of TURKOVAC and two-dose regimen of CoronaVac vaccines for Real Time-PCR confirmed symptomatic COVID-19 disease.

SECONDARY OUTCOMES:
To evaluate the efficacy of one dose of CoronaVac with one dose of TURKOVAC for Real Time-PCR-confirmed symptomatic COVID-19 disease. | after one dose of vaccination
  The protection rate of, at least, one dose of SARS-CoV-2 vaccine against Real Time-PCR confirmed symptomatic COVID-19.
To assess the safety of TURKOVAC and CoronaVac vaccines. | after one dose of vaccination
  The incidence of adverse reactions after one dose of vaccination.
To assess the immunogenicity of TURKOVAC and CoronaVac vaccines. | 14 days after each dose vaccination
  The seroconversion rate, seropositivity rate 14 days after each dose vaccination.
To determine the seropositivity rate of SARS-CoV2 specific binding antibody at 42, 56, 70, 168 and 224 days after the first dose. | at 42, 56, 70, 168 and 224 days after the first dose.
  The seroconversion rate, seropositivity rate at 42, 56, 70, 168 and 224 days after the first dose.
To evaluate SARS-CoV2 neutralizing antibodies by neutralization test on the first dose day and at 42, 56, 70, 168 and 224 days after the first dose among the subjects vaccinated with TURKOVAC and the subjects vaccinated with CoronaVac. | at 42, 56, 70, 168 and 224 days after the first dose
  Geometric mean titer and Geometric mean intensity of neutralizing antibody and immunoglobulin G at 42, 56, 70, 168 and 224 days after the first dose.
To evaluate the efficacy and hospitalization and death rates of two doses of TURKOVAC vaccine against severe cases of COVID-19. | 2 weeks after the second dose of vaccination
  The protection rate of a two-dose of SARS-CoV-2 vaccine against rates of hospitalization, disease severity/and death two weeks after the second dose of vaccination.
To determine the incidence of adverse reactions and serious adverse events. | after one dose of vaccination
  The incidence of adverse reactions within after one dose of vaccination.
To evaluate the SARS-CoV2 protein peptide pool-specific T cells (T cell activation) on the first dose day and at 42, 70, 168 and 224 days after the first dose. | at 42, 70, 168 and 224 days after the first dose
  Geometric mean percentage of SARS-CoV2 protein peptide pool specific T-cell determined by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Durusu Tanrıöver, Prof., Principal Investigator — Faculty Member
Locations (29):
- Turkey (Türkiye) (29):
  - T.R. Ministry of Health Ankara City Hospital, Infectious Diseases and Clinical Microbiology Clinic, Ankara, Turkey Region
  - Çukurova University Faculty of Medicine, Department of Infectious Diseases, Adana
  - Hacettepe University Faculty of Medicine Department of Infections Diseases and Clinical Microbiology, Ankara
  - Ankara University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Ankara
  - Gazi University Faculty of Medicine, Department of Infectious Diseases, Ankara
  - T.R. Ministry of Health Ankara Keçiören Sanatorium Ataturk Chest Diseases and Thoracic Surgery Training and Research Hospital, Ankara
  - T.R. Ministry of Health Ankara Training and Research Hospital Infectious Diseases Clinic, Ankara
  - Akdeniz University Faculty of Medicine, Department of Infectious Diseases, Antalya
  - Uludağ University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Bursa
  - Dicle University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Diyarbakır
  - Gaziantep University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Gaziantep
  - Acıbadem Atakent Hospital, Infectious Diseases and Clinical Microbiology, Istanbul
  - Cerrahpaşa Faculty of Medicine, Department of Internal Medicine - Department of Infectious Diseases and Clinical Microbiology, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Istanbul
  - T.R. Ministry of Health Başakşehir Çam ve Sakura City Hospital, Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Bakirkoy Dr. Sadi Konuk Training and Research Hospital (Yeşilköy Prof.Dr. Murat Dilmener Emergency Hospital), Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Prof. Dr. Cemil Taşçıoğlu City Hospital, Infectious Diseases Clinic, Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital (Prof. Dr. Feriha Öz Emergency Hospital), Istanbul
  - T.R. Ministry of Health İstanbul Şişli Hamidiye Etfal Training and Research Hospital, Clinical Microbiology Clinic, Istanbul
  - University of Health Sciences İstanbul Ümraniye Training and Research Hospital, Istanbul
  - Ege University Faculty of Medicine Hospital, Department of Infectious Diseasesaculty of Medicine Hospital, Department of Infectious Diseases, Izmir
  - T.R. Ministry of Health İzmir Provincial Health Directorate Health Sciences University Dr Suat Seren Chest Diseases And Chest Surgery Training And Research Hospital, Izmir
  - T.R. Ministry of Health İzmir Provincial Health Directorate İzmir Health Sciences University Tepecik Training and Research Hospital, Infectious Diseases, Izmir
  - Erciyes University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Kayseri
  - T.R. Ministry of Health Kayseri City Training and Research Hospital, Infectious Diseases and Clinical Microbiology Department, Kayseri
  - Kocaeli University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Kocaeli
  - Malatya İnönü University Faculty of Medicine, Department of Infectious Diseases, Malatya
  - Ondokuz Mayıs University Istanbul Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Samsun
  - Karadeniz Technical University Medical Faculty Hospital, Department of Infectious Diseases and Clinical Microbiology, Trabzon

REFERENCES:
- [Background] Pavel STI, Yetiskin H, Aydin G, Holyavkin C, Uygut MA, Dursun ZB, Celik I, Cevik C, Ozdarendeli A. Isolation and characterization of severe acute respiratory syndrome coronavirus 2 in Turkey. PLoS One. 2020 Sep 16;15(9):e0238614. doi: 10.1371/journal.pone.0238614. eCollection 2020. PMID 32936826